CLINICAL TRIAL: NCT04749784
Title: Double-blind, Randomised, Placebo-controlled Study to Evaluate the Benefit and Tolerability of Arterin Cholesterol for Reduction of Lipid Levels
Brief Title: Effects of Arterin Cholesterol for Reduction of Lipid Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Perrigo CSCI (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PERI/002620
Record Dates: First submitted 2020-10-28; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Blood Cholesterol Lowers; LDL-C
Keywords: nutritional supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High dose IP (Experimental): Two tablets IP daily for 12 weeks
  Interventions: Dietary Supplement: High Dose Arterin Cholesterol
- Low dose IP (Experimental): One tablet IP + one tablet placebo daily for 12 weeks
  Interventions: Dietary Supplement: Low Dose Arterin Cholesterol
- Placebo (Placebo Comparator): Two tablets placebo daily for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High Dose Arterin Cholesterol — 240mg active ingredient daily
  Arms: High dose IP
Dietary Supplement: Low Dose Arterin Cholesterol — 120mg active ingredient daily
  Arms: Low dose IP
Dietary Supplement: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The main objective of this double-blind, randomised, placebo-controlled study is to assess the benefit and tolerability of Arterin Cholesterol in subjects with elevated lipid levels within a 12-week period of use.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. 18 to 65 years old
3. BMI 25 - 29.9 kg/m2
4. Generally in good health
5. LDL-C level between 3.359-4.884 mmol/L (130-189 mg/dL)
6. Stable body weight for at least 3 months prior to study inclusion (<3 kg weight change) (self-reported)
7. Not smoking, at least 6 months prior to study inclusion and throughout the study
8. Electrocardiogram (ECG) without pathological findings at V1
9. Readiness and ability to comply with study requirements, in particular:

   * to take IP as recommended
   * to avoid the use of any nutritional, medical and further interventional options for reduction/maintenance of lipid levels during the study (other than the IP)
   * to avoid consumption of grapefruit, but otherwise keep the dietary habits
   * to keep the habitual level of physical activity during the study
10. Women of childbearing potential:

    * commitment to use contraception methods
    * negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1
11. Readiness not to participate in another clinical study during this study

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product
2. LDL-C level ≥4.910 mmol/L (≥190 mg/dL)
3. Total cholesterol level ≥7.254 mmol/L (≥280 mg/dL)
4. Triglyceride level ≥2.851 mmol/L (≥250 mg/dL)
5. HDL-C level <1.034 mmol/L (<40 mg/dL)
6. Known genetic hyperlipidemia
7. Known family history of dyslipidemia
8. History and/or presence of clinically significant known (self-reported) condition/disorder, which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

   * cardiovascular disease/disorder (myocardial infarction, angina pectoris, stroke, heart failure, arrhythmia) within 6 months or requiring percutaneous coronary intervention or coronary artery bypass surgery
   * untreated or non-stabilised thyroid gland disorder
   * untreated or non-stabilised hypertension (regular systolic blood pressure

     ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg)
   * acute or chronic gastrointestinal (GI) disease or digestion/absorption disorders (e.g. inflammatory bowel disease, coeliac disease, pancreatitis etc.)
   * untreated/non-stabilised diabetes mellitus type 1 or 2
   * acute or chronic psychotic disorder
   * any other relevant serious diseases
9. Deviation of safety laboratory parameter(s) at V1 that is:

   * clinically significant or
   * >2x upper limit of normal, unless the deviation is justified by a previously known not clinically relevant condition (e.g. Gilbert's syndrome)
10. Regular medication and/or supplementation and/or treatment (including any natural health products) within the last 2 months prior to V1 and during the study, as per investigator judgement:

    * lipid lowering products (known to affect lipid metabolism, platelet function, antioxidant status, etc.), including dietary or health supplements (e.g. omega-3 fatty acids, calcium, oat fiber, niacin, green tea extract, plant sterols, soy protein, psyllium seed husk, probiotics/prebiotics)
    * products that can influence cholesterol levels (e.g. corticosteroids, beta blockers, amiodarone, estrogen, anabolic steroids), unless it is long term and stabilised (contraceptives are allowed in case of a stable continuous intake before and during the study)
    * that could influence gastrointestinal functions (e.g. laxatives, opioids, anticholinergics etc.)
    * any other, which could interfere with the results of the study or the safety of the subject
11. Women of childbearing potential: pregnancy or nursing
12. History of or current abuse of drugs, alcohol or medication
13. Participation in another study during the last 30 days prior to V1
14. Any other reason for exclusion as per investigator's judgment, e.g. insufficient compliance with study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
LDL-C levels between High Dose IP and placebo | 12 weeks
  Difference in LDL-C levels between High Dose IP and placebo at study end compared to baseline

SECONDARY OUTCOMES:
Difference LDL-C levels between Low Dose IP and placebo | 12 weeks
  Difference in change of LDL-C levels between Low Dose IP and placebo at study end compared to baseline
Difference between combined IP vs. placebo | 12 weeks
  Difference in LDL-C levels at V3, V4 and V5 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in change in LDL-C levels at V3, V4 and V5, each in comparison to V2 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in TC levels at V3, V4 and V5 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in change in TC levels at V3, V4 and V5, each in comparison to V2 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in TG levels at V3, V4 and V5 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in change in TG levels at V3, V4 and V5, each in comparison to V2 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in HDL-C levels at V3, V4 and V5 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in change in HDL-C levels at V3, V4 and V5, each in comparison to V2 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in LDL-C/HDL-C ratio at V3, V4 and V5 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in change in LDL-C/HDL-C ratio at V3, V4 and V5, each in comparison to V2 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in SCORE value at V3, V4 and V5 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in change in SCORE value at V3, V4 and V5, each in comparison to V2 between combined IP vs. placebo
Difference between combined IP vs. placebo | 12 weeks
  Difference in global evaluation of benefit by the subject and investigator at study end between combined IP vs. placebo

OTHER OUTCOMES:
Difference in tolerability parameters between groups | 12 weeks
  Changes in safety laboratory parameters at study end in comparison to V1
Difference in tolerability parameters between groups | 12 weeks
  Changes in vital signs throughout the study
Difference in tolerability parameters between groups | 12 weeks
  Assessment of adverse events throughout the study
Difference in tolerability parameters between groups | 12 weeks
  Global evaluation of tolerability by subject and investigator at study end
Difference in body weight between groups | 12 weeks
  Changes in body weight throughout the study
Difference in dietary habits between groups | 12 weeks
  Changes in dietary habits throughout the study
Difference in physical activity between groups | 12 weeks
  Changes in level of physical activity throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, MD, Principal Investigator — Analyze & Realize
Locations (1):
- analyze & realize GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No